CLINICAL TRIAL: NCT02887872
Title: Combining Electrical Stimulation and a Dynamic Hand Orthosis for Functional Recovery in Chronic Stroke
Brief Title: Electrical Stimulation and a Dynamic Orthosis for Stroke Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-020
Record Dates: First submitted 2016-08-16; First posted 2016-09-02 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2016-08

CONDITIONS: Stroke
Keywords: stroke; upper extremity function; rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pilot data (Experimental): Four participants with chronic stroke participated in a 45-minute combined electrical stimulation-dynamic hand orthosis regimen using the affected upper extremity (UE) 5X/week for 6 weeks.
  Interventions: Other: Electrical stimulation-dynamic hand orthosis

INTERVENTIONS:
Other: Electrical stimulation-dynamic hand orthosis — Each participant participated in the electrical stimulation-dynamic hand orthosis regimen. Repetitive grasp/release motions were performed for 30 minutes while wearing the dynamic hand orthosis. This was followed by 15 minutes of electrical stimulation applied to forearm extensor muscles. This regimen was performed daily, 5X/week for 6 weeks.
  Other Names: Empi 300PV neuromuscular electrical stimulation unit; SaeboFlex dynamic hand orthosis

SUMMARY:
Objective: To explore the effectiveness of a combined neuromuscular electrical stimulation (ES) and dynamic hand orthosis (DHO) regimen used with a small group of persons with chronic stroke in improving ability to perform daily tasks. Method: Four participants with chronic stroke participated in the combined ES-DHO regimen using the affected upper extremity (UE) five times (5X) per week for 6 weeks. Outcome measures included grip strength, range of motion (ROM), and analysis of muscle activation/deactivation during release of grasp through electromyography (EMG). Ability to perform daily functional tasks was assessed using the Assessment of Motor and Process Skills (AMPS). Results: Preliminary results suggest that improvements in strength, ROM and grasp deactivation are possible with the combined ES-DHO regimen. Ability to perform daily functional tasks improved in all participants. Conclusion: Results should be interpreted cautiously due to the pilot nature of the study and small participant number. Further research in this area is warranted.

DETAILED DESCRIPTION:
The purpose of this pilot study was to explore the outcomes on performance of functional daily living tasks following a six-week combined regimen using ES and the SaeboFlex orthosis with repetitive task training (RTT) in four persons with chronic stroke. Functional outcomes were assessed before and after (pre-post design) a six-week combined treatment regimen using the DHO during RTT followed by a regimen of ES. Feasibility and logistics for translation of these preliminary results to a larger, more comprehensive controlled trial were explored. Participants donned the orthosis on the affected upper extremity with therapist assistance and performed the RTT grasp/release practice daily for 30 minutes, 5X/week for 6 weeks (30 sessions).Following completion of the grasp/release practice, ES to the finger extensor muscles was provided for 15 minutes. Goniometry to measure range of motion (ROM) at wrist and fingers, dynamometry to measure hand strength, electromyography (EMG) collection to measure muscle activation/deactivation, and AMPS testing to measure functional activity performance were performed before starting the intervention (baseline) and one day after the final training session. Gains in grip strength, 3rd metacarpophalangeal (MP) flexion, AMPS motor score, and improved deactivation of grasp were observed in all participants. Wrist extension, 3rd MP extension, AMPS process score, EMG root mean square (RMS) and time to release grasp improved in three of the four participants.These preliminary pilot results begin to suggest that gains can be made in impairment areas of strength, ROM, and the functional movement pattern of grasp release with a combined ES-DHO program in individuals with chronic stroke. Perhaps most importantly, the results may indicate that this type of training may translate to improvement in performance of daily living tasks. Completion of this work suggests that a larger trial is feasible and logistically able to be performed. The preliminary data are limited in that only four volunteers with chronic stroke were studied, so the small numbers involved restrict generalizations of effectiveness and comprehensive analysis of outcomes.

ELIGIBILITY:
Inclusion Criteria

1. have a diagnosis of ischemic or hemorrhagic stroke that occurred at least six months prior to date of participation;
2. be between 20 and 85 years of age;
3. exhibit a minimal amount of upper extremity movement (approximately 10° active wrist or digit movement);
4. be able to communicate orally and provide informed consent; and
5. be able to comprehend the responsibilities and procedures related to the study.

Exclusion Criteria:

(1) having one or more contraindicated conditions to receive electrical stimulation (implanted pacemaker/electronics, surgical hardware, tumors, cellulitis, open wounds, etc.)

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline performance of functional tasks to post-intervention performance of functional tasks | Before and after 6-week (30 visits) electrical stimulation-dynamic hand orthosis intervention
  Motor and process scores of the Assessment of Motor and Process Skills (AMPS) test

SECONDARY OUTCOMES:
Change from baseline grip strength to post-intervention grip strength | Before and after 6-week (30 visits) electrical stimulation-dynamic hand orthosis intervention
  Strength of grip in affected hand measured through dynamometry
Change from baseline range of motion in wrist and metacarpal joint to post-intervention range of motion in wrist and metacarpal joint | Before and after 6-week (30 visits) electrical stimulation-dynamic hand orthosis intervention
  Range of motion (flexion/extension)of affected wrist and 3rd metacarpal joint measured through goniometry performed by blinded evaluator
Change from baseline forearm muscle activation/deactivation to post-intervention forearm muscle activation/deactivation | Before and after 6-week (30 visits) electrical stimulation-dynamic hand orthosis intervention
  Root mean square and time course of electromyographical (EMG) signal of extensor muscles persisting after auditory cue to release grasp

CONTACTS AND LOCATIONS:
Overall Officials: Barbara M. Doucet, PhD, Principal Investigator — Louisiana State University Health Sciences Center
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Individual data are confidential.

REFERENCES:
- [Result] Aoyagi Y, Tsubahara A. Therapeutic orthosis and electrical stimulation for upper extremity hemiplegia after stroke: a review of effectiveness based on evidence. Top Stroke Rehabil. 2004 Summer;11(3):9-15. doi: 10.1310/6Q5Q-69PU-NLQ9-AVMR. PMID 15480949
- [Result] Barry JG, Ross SA, Woehrle J. Therapy incorporating a dynamic wrist-hand orthosis versus manual assistance in chronic stroke: a pilot study. J Neurol Phys Ther. 2012 Mar;36(1):17-24. doi: 10.1097/NPT.0b013e318246203e. PMID 22354108
- [Result] de Kroon JR, IJzerman MJ. Electrical stimulation of the upper extremity in stroke: cyclic versus EMG-triggered stimulation. Clin Rehabil. 2008 Aug;22(8):690-7. doi: 10.1177/0269215508088984. PMID 18678569
- [Result] Doucet BM, Griffin L. Variable stimulation patterns for poststroke hemiplegia. Muscle Nerve. 2009 Jan;39(1):54-62. doi: 10.1002/mus.21114. PMID 19086075
- [Result] Doucet BM, Lam A, Griffin L. Neuromuscular electrical stimulation for skeletal muscle function. Yale J Biol Med. 2012 Jun;85(2):201-15. Epub 2012 Jun 25. PMID 22737049
- [Result] Hoffman HB, Blakey GL. New design of dynamic orthoses for neurological conditions. NeuroRehabilitation. 2011;28(1):55-61. doi: 10.3233/NRE-2011-0632. PMID 21335678
- [Result] Lee YY, Lin KC, Cheng HJ, Wu CY, Hsieh YW, Chen CK. Effects of combining robot-assisted therapy with neuromuscular electrical stimulation on motor impairment, motor and daily function, and quality of life in patients with chronic stroke: a double-blinded randomized controlled trial. J Neuroeng Rehabil. 2015 Oct 31;12:96. doi: 10.1186/s12984-015-0088-3. PMID 26520398
- [Result] Page SJ, Levin L, Hermann V, Dunning K, Levine P. Longer versus shorter daily durations of electrical stimulation during task-specific practice in moderately impaired stroke. Arch Phys Med Rehabil. 2012 Feb;93(2):200-6. doi: 10.1016/j.apmr.2011.09.016. PMID 22289227
- [Result] Persch AC, Page SJ, Murray C. Paretic upper extremity movement gains are retained 3 months after training with an electrical stimulation neuroprosthesis. Arch Phys Med Rehabil. 2012 Nov;93(11):2122-5. doi: 10.1016/j.apmr.2012.06.006. Epub 2012 Jun 20. PMID 22728015
- [Result] Quandt F, Hummel FC. The influence of functional electrical stimulation on hand motor recovery in stroke patients: a review. Exp Transl Stroke Med. 2014 Aug 21;6:9. doi: 10.1186/2040-7378-6-9. eCollection 2014. PMID 25276333
- [Result] Singer BJ, Vallence AM, Cleary S, Cooper I, Loftus AM. The effect of EMG triggered electrical stimulation plus task practice on arm function in chronic stroke patients with moderate-severe arm deficits. Restor Neurol Neurosci. 2013;31(6):681-91. doi: 10.3233/RNN-130319. PMID 23963340
- [Result] Sullivan J, Girardi M, Hensley M, Rohaus J, Schewe C, Whittey C, Hansen P, Muir K. Improving arm function in chronic stroke: a pilot study of sensory amplitude electrical stimulation via glove electrode during task-specific training. Top Stroke Rehabil. 2015 Jun;22(3):169-75. doi: 10.1179/1074935714Z.0000000007. Epub 2015 Jan 26. PMID 26084321
- [Result] Sun Y, Boots J, Zehr EP. The lingering effects of a busted myth--false time limits in stroke rehabilitation. Appl Physiol Nutr Metab. 2015 Aug;40(8):858-61. doi: 10.1139/apnm-2014-0523. PMID 26244605
- [Result] Woo Y, Jeon H, Hwang S, Choi B, Lee J. Kinematics variations after spring-assisted orthosis training in persons with stroke. Prosthet Orthot Int. 2013 Aug;37(4):311-6. doi: 10.1177/0309364612461050. Epub 2012 Oct 30. PMID 23112278